CLINICAL TRIAL: NCT03601377
Title: Attention Bias Modification Treatment in Social Anxiety: Avoidance or Exposure to Threatening Faces? The Role of Pre-existing Attentional Biases and State Anxiety
Brief Title: Attention Bias Modification Treatment in Social Anxiety
Acronym: ABMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Collaborators: Youth Board of Cyprus (Unknown); Tel Aviv University (Other)
Responsible Party: Principal Investigator, Klavdia Neophytou, PhD Clinical Psychology Student, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABMT University of Cyprus
Record Dates: First submitted 2018-06-06; First posted 2018-07-26 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Social Anxiety
Keywords: attention bias; treatment predictors

STUDY DESIGN:
Intervention Model Description: Experiment 1: 2 groups (1 intervention and 1 placebo) receive treatment in parallel Experiment 2: 3 groups (2 types of intervention and 1 placebo) receive treatment in parallel
Who Masked: Participant, Investigator
Masking Description: Participants and investigators were blind with regards to which group participants were allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training away from threat (Experimental): Experiment 1 and 2: In the intervention group -training away from threat-, in all angry-neutral faces presentation the probe is presented only after neutral face. Probe type (< or >) is not factorially counterbalanced but there is equal possibility of presentation for each of the following: angry-face location, probe location, or actor.
  Experiment 1: received 8 times (2 times per week for 4 weeks) Experiment 2: received 4 times (2 times for 2 weeks)
  Interventions: Behavioral: Training away from threat
- Training towards threat (Experimental): Only for Experiment 2: The second ABMT condition -training towards threat- is identical to the first one with the exception that in all angry-neutral face presentations the symbol is presented only after threat face. In addition, at the beginning of every session participants will be informed that a random number of participants will have to repeat their speech. They will also be informed that this instruction will be given right after the dot probe task completion. This will be done in order for the participants to maintain their state anxiety but repetition of the speech task will not actually happen at this stage.
  Experiment 2: received 4 times (2 times for 2 weeks)
  Interventions: Behavioral: Training towards threat
- Placebo (Placebo Comparator): Experiment 1 and 2: In the placebo group, angry-face location, probe location and actor are fully counterbalanced with regards to their presentation.
  Experiment 1: received 8 times (2 times per week for 4 weeks) Experiment 2: received 4 times (2 times for 2 weeks)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Training away from threat — Dot-probe task: Pairs of stimuli, angry - neutral face or neutral - neutral faces of the same actor (20 different individuals;10 male, 10 female) are presented horizontally in the centre of the screen (160 trials; 120 angry-neutral and 40 neutral-neutral). Each trial begins with a fixation cross (500 ms), on which the participants are instructed to focus their gaze. After that a pair of faces follows which is presented on the screen for 500ms. After the faces presentation a small visual probe (< or >) appears at the same place of one of the two faces. Participants have to determine which symbol appeared by clicking right or left on the mouse as quickly as possible. The target probe remains on the screen until there is a response, which starts a new trial.
  Arms: Training away from threat
Behavioral: Training towards threat — Dot-probe task: Pairs of stimuli, angry - neutral face or neutral - neutral faces of the same actor (20 different individuals;10 male, 10 female) are presented horizontally in the centre of the screen (160 trials; 120 angry-neutral and 40 neutral-neutral). Each trial begins with a fixation cross (500 ms), on which the participants are instructed to focus their gaze. After that a pair of faces follows which is presented on the screen for 500ms. After the faces presentation a small visual probe (< or >) appears at the same place of one of the two faces. Participants have to determine which symbol appeared by clicking right or left on the mouse as quickly as possible. The target probe remains on the screen until there is a response, which starts a new trial.
  Arms: Training towards threat
Behavioral: Placebo — Dot-probe task: Pairs of stimuli, angry - neutral face or neutral - neutral faces of the same actor (20 different individuals;10 male, 10 female) are presented horizontally in the centre of the screen (160 trials; 120 angry-neutral and 40 neutral-neutral). Each trial begins with a fixation cross (500 ms), on which the participants are instructed to focus their gaze. After that a pair of faces follows which is presented on the screen for 500ms. After the faces presentation a small visual probe (< or >) appears at the same place of one of the two faces. Participants have to determine which symbol appeared by clicking right or left on the mouse as quickly as possible. The target probe remains on the screen until there is a response, which starts a new trial.
  Arms: Placebo

SUMMARY:
This study evaluates attention modification in social anxiety and It is comprised by 2 experiments. At experiment 1 socially anxious participants will receive either training away from threatening faces or placebo intervention and at experiment 2 they will receive either one of these 2 groups or training towards threatening faces. At experiment 2 training will be done under state anxiety levels (video-recording of a speech). Anxiety levels (self-reports, physiological and behavioral measures) as well as attentional biases changes will be examined at pre and post - intervention levels plus 6 months follow-up only for experiment 1.

DETAILED DESCRIPTION:
Social anxiety is a highly prevalent disorder in the population. Even though there are effective interventions that can help people who suffer from it, many of them do not seek or receive an evidence-based, face to face treatment. According to cognitive models, attention to social threat is one of the principles that maintain social anxiety. In fact, individuals with social anxiety present attention bias to threat stimuli. However, there is inconsistency in the literature with regards to attentional biases that individuals with anxiety present. A recent model is the vigilance-avoidance hypothesis, in which socially anxious initially focus on the threat and then they avoid it. Therefore, better understanding and then aiming to modify these attentional biases in a computerized manner, with minimal therapist interaction can be a novel and promising way to treat social anxiety, even among patients who avoid presenting for therapy.

Two experiments are aiming to shed some light with regards to the effect of attention bias modification treatment in individuals with social anxiety, taking into consideration the previous mixed results. The first experiment compares training attention to be directed away from threat with a placebo treatment. Approximately 60 socially anxious individuals are randomly allocated in the 2 groups. A structured interview and self-report assessment are done pre-treatment, post-treatment and 6 months follow-up.

The second experiment adds a third group of training towards threat (i.e. exposure), investigating if changing attentional avoidance can also affect anxiety levels. Moreover, the second experiment attempts to improve the typical attention modification paradigm by targeting treatment to participants' identified pre-experimental attentional biases. In addition, predictors of treatment effectiveness will be studied and particularly pre-intervention attentional biases as well as state anxiety. Participants are approximately 90 adults with social phobia who are randomly allocated in treatment and placebo groups. In experiment 2 participants will also be assessed behaviourally as well as physiologically to better demonstrate that anxiety reactions to anxiogenic situations have been reduced between pre and post treatment and that they are smaller than those of a placebo control group.

It is expected that participants in the intervention groups will show reduced attentional bias and social anxiety symptoms in comparison with the placebo group in both studies. In addition, the kind of pre-intervention bias as well as state anxiety will moderate anxiety changes. This study will enrich existing research on attention bias modification treatment by shedding light into potential mechanisms of change and will examine ways to improve the efficacy of this intervention.

ELIGIBILITY:
Inclusion Criteria:

1) highly socially anxious students (based on self-report questionnaire)

Exclusion Criteria:

1. suicidal intent,
2. substance abuse,
3. primary diagnosis of post-traumatic stress disorder, obsessive-compulsive disorder,
4. or past schizophrenia, bipolar disorder, organic mental disorder,
5. any concurrent psychotherapy,
6. changes in medication during the 12 weeks prior to study and
7. CBT therapy 6 months before the beginning of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Social Anxiety levels | Pre-treatment (day 1)
  Experiment 1 & 2: self-reported questionnaires, with the primary one to be Social Phobia and Anxiety Inventory-23.
Social Anxiety changes | Experiment 1: 4 weeks after the day 1, Experiment 2: 3 weeks after the day 1 (Post-treatment)
  Experiment 1 & 2: Measured in self-reported questionnaires with the primary one to be Social Phobia and Anxiety Inventory-23.
Social Anxiety changes | 6 months after day 1 (Follow-up)
  Only for experiment 1: Measured in self-reported questionnaires with the primary one to be Social Phobia and Anxiety Inventory-23.
Attentional Biases | Pre-treatment (day 1)
  For experiment 1: Assess kind of attentional biases using the dot-probe task (comparison of reaction time to threatening and a neutral stimulus).
  For experiment 2: Assess kind of attentional biases using the eye-tracking task (measuring eye gaze).
Attentional Biases changes | 4 weeks after the day 1 (Post-treatment)
  For experiment 1: Assess kind of attentional biases using the dot-probe task (comparison of reaction time to threatening and a neutral stimulus).
  For experiment 2: Assess kind of attentional biases using the eye-tracking task (measuring eye gaze).
Attentional Biases changes | 6 months after day 1 (Follow-up)
  Only for experiment 1: Assess kind of attentional biases using the dot-probe task (comparison of reaction time to threatening and a neutral stimulus).
Physical social anxiety levels | Pre-treatment (day 1)
  Only for experiment 2: measured through physiological measures, with the primary one to be heart rate.
Physical social anxiety changes | 3 weeks after the day 1 (Post-treatment)
  Only for experiment 2: measured through physiological measures, with the primary one to be heart rate.

SECONDARY OUTCOMES:
Social Anxiety levels (clinical interview) | Pre-treatment (day 1)
  Experiment 1 & 2: measured through clinical interview, Anxiety Disorders Interview Schedule (ADIS) adult version.
Physical social anxiety levels 1 | Pre-treatment (day 1)
  Only for experiment 2: measured through skin conductance
Physical social anxiety levels 2 | Pre-treatment (day 1)
  Only for experiment 2: measured through corrugator supercilii
Social anxiety changes | 4 weeks after the day 1 (Post-treatment)
  Experiment 1: measured through clinical interview, Anxiety Disorders Interview Schedule (ADIS) adult version.
Physical social anxiety changes 1 | 3 weeks after the day 1 (Post-treatment)
  Only for experiment 2: measured through skin conductance
Social anxiety changes | 6 months after day 1 (follow-up)
  Experiment 1: measured through clinical interview, Anxiety Disorders Interview Schedule (ADIS) adult version.
Physical social anxiety changes 2 | 3 weeks after the day 1 (Post-treatment)
  Only for experiment 2: measured through corrugator supercilii

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Panayiotou, PhD, Study Director — Associate Prof., Department of Psychology, University of Cyprus
Locations (1):
- Department of Psychology, University of Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amir N, Beard C, Taylor CT, Klumpp H, Elias J, Burns M, Chen X. Attention training in individuals with generalized social phobia: A randomized controlled trial. J Consult Clin Psychol. 2009 Oct;77(5):961-973. doi: 10.1037/a0016685. PMID 19803575
- [Background] Bar-Haim Y. Research review: Attention bias modification (ABM): a novel treatment for anxiety disorders. J Child Psychol Psychiatry. 2010 Aug;51(8):859-70. doi: 10.1111/j.1469-7610.2010.02251.x. Epub 2010 May 6. PMID 20456540